CLINICAL TRIAL: NCT02669849
Title: A Phase 2b/3, Double-blind, Randomized, Placebo Controlled, Multicenter Study to Assess the Efficacy and Safety of VX-210 in Subjects With Acute Traumatic Cervical Spinal Cord Injury
Brief Title: Study to Assess the Efficacy and Safety of VX-210 in Subjects With Acute Traumatic Cervical Spinal Cord Injury
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX15-210-101
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Cervical Spinal Cord Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- VX-210 (Experimental)
  Interventions: Drug: VX-210

INTERVENTIONS:
Drug: VX-210
  Arms: VX-210
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of VX-210 in subjects with Acute Traumatic Cervical Spinal Cord Injury. Secondary objectives include the specific evaluation of the effects of VX-210 on neurological recovery and daily function after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Acute traumatic cervical SCI, motor level of C4, C5, C6, or C7 on each side:

  * Screening UEMS score must be ≤16 points on each side.
  * AIS A subjects with a C4 motor level on both sides must have at least 1 point of motor activity between C5 and T1 on at least 1 side.
  * AIS B subjects with a C4 motor level on both sides must have at least 1 point of motor activity between C5 and C7 on at least 1 side.
* American Spinal Injury Association Impairment Scale (AIS) grade A or AIS grade B.
* Scheduled and planned to undergo a spinal decompression/stabilization surgery that commences within 72 hours after the initial injury.
* Computed tomography (CT) scan or magnetic resonance imaging (MRI) is consistent with the subject's neurological deficit.

Exclusion Criteria:

* Participation in any other clinical study for acute SCI without approval by the sponsor.
* Inability to undergo decompression/stabilization surgery that commences within 72 hours after injury.
* One or more upper extremity muscle groups untestable during screening ISNCSCI examination.
* Acute SCI from gunshot or penetrating/stab wound; non-traumatic SCI (e.g., transverse myelitis, acute disc herniation); brachial plexus injury; complete spinal cord transection; or multifocal SCI.
* Females who are breastfeeding or have a positive serum pregnancy test.
* Body mass index (BMI) of ≥40 kg/m^2 at screening.
* History of an adverse reaction to a fibrin sealant or its components.
* Unconsciousness or other mental impairment that precludes reliable International Standards for the Neurological Classification of Spinal Cord Injury (ISNCSCI) examination.
* Known immunodeficiency, including human immunodeficiency virus, or use of immunosuppressive or cancer chemotherapeutic drugs.
* Any significant medical or psychiatric comorbidities that would significantly increase the risk of study enrollment and/or significantly interfere with study outcomes or assessments, in the judgment of the investigator.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (33):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Fresno, California
  - Orange, California
  - Sacramento, California
  - Jacksonville, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Falls Church, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Seattle, Washington
- Canada (6):
  - Vancouver, British Colombia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to receive a single 9-mg dose of VX-210 or a placebo (buffer solution). A single 3-mg dose of VX-210 in fibrin sealant was initially included but was subsequently removed during the study through a protocol amendment. The 3-mg arm was not analyzed for primary and secondary efficacy and pharmacokinetic analysis.
Pre-assignment Details: A total of 70 participants were randomized, out of which 67 participants received the study drug.
Groups:
- Placebo: Participants who received placebo matched to VX-210 as a single dose in fibrin sealant topically to the dural surface of the spinal cord within 72 hours after the initial injury.
- VX-210 3 mg: Participants who received VX-210 3 milligram (mg) as a single dose in fibrin sealant topically to the dural surface of the spinal cord within 72 hours after the initial injury.
- VX-210 9 mg: Participants who received VX-210 9 mg as a single dose in fibrin sealant topically to the dural surface of the spinal cord within 72 hours after the initial injury.
Period: Overall Study
Arm/Group | Placebo | VX-210 3 mg | VX-210 9 mg
Started | 29 | 6 | 32
Completed | 11 | 4 | 8
Not Completed | 18 | 2 | 24
Not completed — Withdrawal of Consent (not due to AE) | 0 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 3
Not completed — Death | 1 | 1 | 2
Not completed — Study terminated by sponsor | 16 | 1 | 14
Not completed — Other | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Overall number of Baseline participants includes all randomized participants who received study drug.
Groups:
- VX-210 3 mg: Participants who received VX-210 3 mg as a single dose in fibrin sealant topically to the dural surface of the spinal cord within 72 hours after the initial injury.
- Total: Total of all reporting groups
Arm/Group | Placebo | VX-210 3 mg | VX-210 9 mg | Total
Number analyzed (Participants) | 29 | 6 | 32 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (17.4) | 39.5 (24.4) | 43.4 (17.3) | 43.2 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 6 | 16
  Male | 21 | 4 | 26 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 28 | 5 | 31 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 2 | 0 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 0 | 5 | 11
  White | 19 | 3 | 21 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 1 | 5
Upper Extremity Motor Score (UEMS) [Mean (Standard Deviation); unit: units on a scale] — UEMS focuses selectively on the hand and arm control most relevant to individuals with a cervical spinal cord injury. UEMS ranges from 0 to 50, where highest score indicates the positive movement of hand and arm.
  units on a scale | 13.00 (8.96) | 10.17 (6.59) | 14.03 (8.33) | 13.24 (8.43)

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper Extremity Motor Score (UEMS)
Description: UEMS focuses selectively on the hand and arm control most relevant to individuals with a cervical spinal cord injury. UEMS ranges from 0 to 50, where a higher score indicates a better movement of hand and arm.
Time Frame: From baseline at 6 months post-treatment
Population: The "Overall Number of Participants Analyzed" included all randomized subjects who received study drug. As per the amended protocol, the 3 mg arm was no longer planned to be assessed for any primary or secondary outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VX-210 9 mg
Number analyzed (Participants) | 29 | 32
units on a scale | 8.90 (9.48) | 8.69 (7.35)
Statistical Analysis 1: Comparison: Placebo vs VX-210 9 mg; Test type: Superiority; p = 0.7519, Mixed-effects model for repeated measure; Least Squares (LS) Mean Difference = -0.69, 95% CI 2-sided [-5.08 to 3.69]

2. Secondary Outcome: Spinal Cord Independence Measure (SCIM) III Self-Care Subscore
Description: SCIM self-care subscore measures self-care abilities (feeding, dressing, grooming, bathing), respiration and sphincter management and mobility. The score ranges from 0-20, where a higher score represents a better outcome.
Time Frame: At 6 months post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VX-210 9 mg
Number analyzed (Participants) | 29 | 32
units on a scale | 6.2 (7.0) | 5.9 (6.6)

3. Secondary Outcome: Capabilities of Upper Extremity Test (CUE-T) Score
Description: CUE-T measures a participant's ability to perform specific functional movements/tasks with the arms and hands (for example: grasping a pencil, pushing or lifting a weight). CUE-T score ranges from 0-128, where a higher score indicates an improvement in participant's ability.
Time Frame: At 6 months post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VX-210 9 mg
Number analyzed (Participants) | 29 | 32
units on a scale | 39.6 (38.4) | 42.8 (41.1)

4. Secondary Outcome: Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) Quantitative Prehension Score
Description: GRASSP measures participant's ability to perform specific functional tasks with the arms, hands, and fingers. GRASSP quantitative prehension score ranges from 0-60, where a higher score indicates a better performance.
Time Frame: At 6 months post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | VX-210 9 mg
Number analyzed (Participants) | 29 | 32
units on a scale | 18.9 (19.4) | 20.1 (21.6)

5. Secondary Outcome: Percentage of American Spinal Injury Association Impairment Scale (AIS) Grade Responders
Description: AIS ranks impairment according to body-wide motor/sensory results: Grade A: Complete (no sensory or motor function is preserved in the sacral segments S4 to 5); Grade B: Sensory Incomplete (sensory but not motor function is preserved below the neurological level and includes the sacral segments S4 to 5); Grade C: Motor Incomplete (motor function is preserved at the most caudal sacral segments); Grade D: Motor Incomplete (motor incomplete status as defined above, with at least half or more of key muscle functions below the single neurological level of injury having a muscle grade >=3; Grade E: Normal (sensation and motor function as tested are graded as normal in all segments). An AIS responder was defined as a subject with improvement by ≥2 AIS grades (i.e., baseline AIS Grade A changed to Grade C, D, or E; baseline AIS Grade B changed to D or E at 6 months after treatment).
Time Frame: At 6 months post-treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VX-210 9 mg
Number analyzed (Participants) | 29 | 32
percentage of participants | 30.0 | 26.7

6. Secondary Outcome: Percentage of Motor Level Responders
Description: The motor level score for the right or left side assesses contraction strength of 10 key muscles in the upper and lower extremities on each side of the body; each muscle receives a score from 0 (total paralysis) to 5 ([normal] active movement). A motor level responder was defined as a subject with improvement by ≥2 motor levels on either side of the body (i.e., baseline level C4 changed to C6, C7, C8 on the left; or baseline level C5 changed to C7, C8 on the right).
Time Frame: At 6 months post-treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | VX-210 9 mg
Number analyzed (Participants) | 29 | 32
percentage of participants | 35.0 | 33.3

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of VX-210
Time Frame: up to 53 hours post-treatment
Population: Pharmacokinetic analysis set included all participants for which PK data was collected. As per the amended protocol, the 3 mg arm was no longer planned to be assessed for any primary or secondary outcome measure.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | VX-210 9 mg
Number analyzed (Participants) | 28
hours (h) | 4.59 [2.58 to 52.38]

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of VX-210
Time Frame: up to 53 hours post-treatment
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | VX-210 9 mg
Number analyzed (Participants) | 28
nanogram per milliliter (ng/mL) | 2.856 (200.35)

9. Secondary Outcome: Area Under Plasma Concentration Time Curve (AUC) of VX-210
Time Frame: up to 53 hours post-treatment
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | VX-210 9 mg
Number analyzed (Participants) | 28
h*ng/mL | 44.683 (284.95)

ADVERSE EVENTS:
Time Frame: Up to 28 months
Description: Death reported under placebo arm was not treatment-emergent.
Arm/Group | Placebo | VX-210 3 mg | VX-210 9 mg
All-Cause Mortality (participants affected / at risk) | 1/29 | 1/6 | 2/32
Serious Adverse Events (participants affected / at risk) | 18/29 | 6/6 | 16/32
Other Adverse Events (participants affected / at risk) | 28/29 | 6/6 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | VX-210 3 mg (N=6) | VX-210 9 mg (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 1
Empyema (Infections and infestations) | 0 | 0 | 1
Haemophilus infection (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 0 | 2
Pneumonia (Infections and infestations) | 4 | 3 | 4
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 0 | 4
Septic shock (Infections and infestations) | 1 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 0 | 1
Autonomic dysreflexia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Neurogenic shock (Vascular disorders) | 0 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | VX-210 3 mg (N=6) | VX-210 9 mg (N=32)
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 6
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 6 | 0 | 4
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 6
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 4 | 0 | 3
Melaena (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 3 | 5
Neurogenic bowel (Gastrointestinal disorders) | 3 | 0 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 2
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 3
Impaired healing (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0
Pain (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 13 | 3 | 16
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 3 | 1 | 0
Infected skin ulcer (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 2
Oral candidiasis (Infections and infestations) | 2 | 1 | 5
Pneumonia (Infections and infestations) | 7 | 2 | 11
Staphylococcal infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 18 | 4 | 18
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1 | 0
Autonomic dysreflexia (Injury, poisoning and procedural complications) | 3 | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Weaning failure (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0
Blood magnesium decreased (Investigations) | 2 | 0 | 2
Blood phosphorus decreased (Investigations) | 1 | 0 | 2
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Haemophilus test positive (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 4 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 3 | 14
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 4
Muscle spasticity (Nervous system disorders) | 2 | 1 | 4
Neuralgia (Nervous system disorders) | 7 | 2 | 10
Nystagmus (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 2 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 1 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 6 | 1 | 9
Delirium (Psychiatric disorders) | 3 | 0 | 2
Depression (Psychiatric disorders) | 7 | 1 | 6
Hallucination (Psychiatric disorders) | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 11 | 2 | 9
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1
Neurogenic bladder (Renal and urinary disorders) | 5 | 0 | 8
Urinary retention (Renal and urinary disorders) | 3 | 1 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 11 | 3 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 3
Deep vein thrombosis (Vascular disorders) | 5 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 10 | 0 | 11
Orthostatic hypotension (Vascular disorders) | 2 | 3 | 5
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT02669849/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02669849/SAP_001.pdf